CLINICAL TRIAL: NCT04837326
Title: Effect of Using White Noise, Embracing and Facilitated Tucking on Physiological Parameters, Crying Duration and Pain During Heel Lance Blood Sampling in Newborns: Randomized Controlled Trial
Brief Title: Effect of Using White Noise, Embracing and Facilitated Tucking in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilekkucu Kalemdar, Associate Prof. Dr, Ordu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24237859-714
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This randomized-controlled experimental study was performed to evaluate the effect of white noise, embracing and facilitated tucking on pain during heel lance blood sampling in newborns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heel Lance Blood Sampling in Facilitated Tucking Position (Experimental): The infants were put in facilitated tucking position by an experienced newborn nurse. They were put in facilitated tucking position so that their arms and legs were in a flexed midline position close to their trunk in a side-lying position. They were positioned so that they could move their extremities freely. They were held in facilitated tucking position for 120 seconds before the procedure. They were kept in facilitated tucking position until the blood sample was taken from the right heel using a lancet. They were released 60 seconds after the procedure and monitored for 120 seconds. The blood samples were taken by the researcher after inserting the lancet in the first try.
  Interventions: Other: Heel Lance Blood Sampling in Facilitated Tucking Position
- Heel Lance Blood Sampling When the Infant is Embraced by the Mother (Experimental): The mother, whose privacy was protected, embraced the infant for 120 seconds before the procedure. The infant was embraced by the mother during the heel lance blood sampling from the left heel using a lancet. They were released 60 seconds after the procedure and monitored for 120 seconds. The blood samples were taken by the researcher after inserting the lancet in the first try.
  Interventions: Other: Heel Lance Blood Sampling When the Infant is Embraced by the Mother
- Heel Lance Blood Sampling Using White Noise (Experimental): The 'Don't Let Your Baby Cry, PT.2' track from the 'Colic' album by Orhan Osman using the 'The Happiest Baby' album by Dr. Harvery Karp which was composed only of intrauterine was made listened to the infants via Xperia Ultra Mp3 Player for 120 seconds before and 120 seconds after the heel lance blood sampling procedure. While white noise was made listened to the infants before, during and after the procedure, Digital Sound LeverMeter brand noise measurement device was put at a distance of 50 cm from the infant and the ambient noise level was adjusted as 55 dB. The blood samples were taken by the researcher after inserting the lancet in the first try.
  Interventions: Other: Heel Lance Blood Sampling Using White Noise
- Control Group (No Intervention): Suitable environmental conditions (ambient temperature, silent environment, etc.) were ensured in the study room for the infant's comfort. A saturation probe was inserted to the right wrist of the infant to monitor him/her. A video record was taken for 120 seconds without any intervention to the infants before and after the heel lance blood sampling procedure. The blood samples were taken by the researcher after inserting the lancet in the first try. Heel lance was performed in clinical routine for preterm infants in the control group.

INTERVENTIONS:
Other: Heel Lance Blood Sampling in Facilitated Tucking Position
  Arms: Heel Lance Blood Sampling in Facilitated Tucking Position
Other: Heel Lance Blood Sampling When the Infant is Embraced by the Mother
  Arms: Heel Lance Blood Sampling When the Infant is Embraced by the Mother
Other: Heel Lance Blood Sampling Using White Noise
  Arms: Heel Lance Blood Sampling Using White Noise

SUMMARY:
This study was conducted to evaluate the effect of using white noise, embracing and facilitated tucking on physiological parameters, crying duration and pain during heel lance blood sampling in healthy newborns.

This study was a prospective, randomized controlled trial. The study was conducted with healthy newborns who were born between 38 and 42 weeks of gestation. The newborns were divided into 4 groups by the applied pain relief methods during heel lance blood sampling in newborns; embracing(n=40), white noise(n=40), facilitated tucking(n=40) and control group (n=40). The physiological changes were evaluated before and after the procedure. NIPS (Neonatal Infant Pain Scale) was used for pain scoring.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of white noise, embracing and facilitated tucking on pain during heel lance blood sampling in newborns.

METHODS This randomized-controlled experimental study was performed to evaluate the effect of white noise, embracing and facilitated tucking on pain during heel lance blood sampling in newborns.

Setting and sample:

The study sample consisted of healthy newborns who were born and monitored in the Neonatology Unit of a university hospital. The sample inclusion criteria were gestational age between 38 and 42 weeks, birth weight of 2500 - 4000 g, Apgar score of 8 and higher at 1st and 5th minute, having breastfed at least half an hour before the procedure, not showing any disease symptom, not having congenital anomaly, getting a good hearing test result and not having received any invasive intervention other than Vitamin K and Hepatitis B vaccine.

Sample size:

Following previous studies, G*Power (v3.1.9.2) was deployed to determine the sample number. According to Jacob Cohen's effect size coefficients, assuming that evaluations carried out among four independent groups would have a large effect size (d=0.40), it was determined that the groups should comprise least 40 people, with a total of 160, for levels of α=0.05 and 1-β=0.95 (80% power). Children were assigned to 4 subgroups through randomization performed using a computer program (www.randomizer.org): group 1 was the control group children who received no intervention for pain relief (n = 40); group 2 received facilitated tucking (n = 40); group 3 received embracing (n = 40); and group 4 received white noise (n = 40).

Intervention:

The mothers were informed by the researcher about the purpose of the study before collecting data. The infants were held by their mothers so that their faces, arms, legs and respirations could be easily viewed by the camera to evaluate the NIPS. All heel lance procedures were performed by the same nurse working on the day shift (who had 6-year NICU experience). The heel lance blood sampling point (outer side of the left heel), the lancet used in the procedure, the sampling technique, and the antiseptic solution (70% alcohol) used in for the procedure were the same for all the groups. The heel lance blood sampling procedure was performed by the researcher in the blood sampling room in the Neonatology ward. Suitable environmental conditions (ambient temperature, silent environment, etc.) were ensured in the study room for the infant's comfort. A saturation probe was inserted to the right wrist of the infant to monitor him/her. The behavioral responses to pain and crying durations of all the responses were recorded by camera before, during and after the procedure. Then, these records were played and the NIPS scores and crying durations of the infants were evaluated. The physiological changes were recorded before, during and after the procedure, respectively. In the data collection stage, 3 persons (nurse putting the infant in facilitated tucking position, nurse taking blood sample, researcher shooting video) were required for facilitated tucking position; 2 persons (nurse taking blood sample and researcher shooting video) for maternal embracing since the infant was held by the mother and 2 persons (nurse taking blood sample and researcher shooting video) for white noise.

Heel Lance Blood Sampling in Facilitated Tucking Position:

The infants were put in facilitated tucking position by an experienced newborn nurse. They were put in facilitated tucking position so that their arms and legs were in a flexed midline position close to their trunk in a side-lying position. They were positioned so that they could move their extremities freely. They were held in facilitated tucking position for 120 seconds before the procedure. They were kept in facilitated tucking position until the blood sample was taken from the right heel using a lancet. They were released 60 seconds after the procedure and monitored for 120 seconds. The blood samples were taken by the researcher after inserting the lancet in the first try.

Heel Lance Blood Sampling When the Infant is Embraced by the Mother:

The mother, whose privacy was protected, embraced the infant for 120 seconds before the procedure. The infant was embraced by the mother during the heel lance blood sampling from the left heel using a lancet. They were released 60 seconds after the procedure and monitored for 120 seconds. The blood samples were taken by the researcher after inserting the lancet in the first try.

Heel Lance Blood Sampling Using White Noise:

The 'Don't Let Your Baby Cry, PT.2' track from the 'Colic' album by Orhan Osman using the 'The Happiest Baby' album by Dr. Harvery Karp which was composed only of intrauterine was made listened to the infants via Xperia Ultra Mp3 Player for 120 seconds before and 120 seconds after the heel lance blood sampling procedure. While white noise was made listened to the infants before, during and after the procedure, Digital Sound LeverMeter brand noise measurement device was put at a distance of 50 cm from the infant and the ambient noise level was adjusted as 55 dB. The blood samples were taken by the researcher after inserting the lancet in the first try.

Control Group:

Suitable environmental conditions (ambient temperature, silent environment, etc.) were ensured in the study room for the infant's comfort. A saturation probe was inserted to the right wrist of the infant to monitor him/her. A video record was taken for 120 seconds without any intervention to the infants before and after the heel lance blood sampling procedure. The blood samples were taken by the researcher after inserting the lancet in the first try. Heel lance was performed in clinical routine for preterm infants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 38 and 42 weeks,
* birth weight of 2500 - 4000 g,
* Apgar score of 8 and higher at 1st and 5th minute,
* having breastfed at least half an hour before the procedure,
* not showing any disease symptom,

Exclusion Criteria:

* having congenital anomaly,
* getting a good hearing test result
* having received any invasive intervention other than Vitamin K and Hepatitis B vaccine.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain | 15 minutes
  Neonatal Infant Pain Scale
Crying Duration | 15 minutes
  Crying durations of the infants.
Physiological Parameters 1 | 15 minutes
  Pulse rate
Physiological Parameters 2 | 15 minutes
  SpO2
Physiological Parameters 3 | 15 minutes
  Respiration rate

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz ÖZORAN, Professor, Study Director — Avrasya University

IPD SHARING:
Plan to Share IPD: No
Results